CLINICAL TRIAL: NCT02302456
Title: Tranexamic Acid for Preventing Postpartum Haemorrhage Following a Vaginal Delivery: a Multicenter Randomised Double Blind Placebo Controlled Trial
Brief Title: Tranexamic Acid for Preventing Postpartum Haemorrhage Following a Vaginal Delivery
Acronym: TRAAP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PHRC 2013-01
Record Dates: First submitted 2014-11-17; First posted 2014-11-27 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Immediate Postpartum Hemorrhage
Keywords: Immediate postpartum hemorrhage; tranexamic acid; prevention
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TXA (Experimental): Intravenous administration of 1g of tranexamic acid within 2 minutes after birth and prophylactic oxytocin administration
  Interventions: Drug: Tranexamic Acid
- Placebo (Placebo Comparator): Intravenous administration of placebo within 2 minutes after birth and prophylactic oxytocin administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic Acid — Intravenous administration of a 10 mL solution containing 1g of tranexamic acid within 2 minutes of birth and routine prophylactic IV injection of oxytocin
  Arms: TXA
Drug: Placebo — Intravenous administration of 10 mL of 0.9% sodium chloride solution within 2 minutes of birth and routine prophylactic IV injection of oxytocin
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess whether the administration of a low dose of tranexamic acid just after vaginal delivery can reduce the incidence of immediate postpartum hemorrhage, in women who receive a prophylactic administration of oxytocin.

DETAILED DESCRIPTION:
Postpartum hemorrhage (PPH) is a major cause of maternal mortality, accounting for one quarter of all maternal deaths worldwide. Its incidence estimates in the literature vary widely, from 3% to 15% of deliveries. Uterotonics after birth are the only intervention that has been shown to be effective for PPH prevention. Tranexamic acid (TXA), an antifibrinolytic agent, has therefore been investigated as a potentially useful complement to uterotonics for prevention because it has been proved to reduce blood loss in elective surgery, bleeding in trauma patients, and menstrual blood loss. Randomized controlled trials for PPH prevention after cesarean (n=10) and vaginal (n=2) deliveries showed that women who had received TXA had a significantly lesser amount of postpartum blood loss without any increase in severe maternal adverse effect. However, overall, the quality of these trials was poor, and they were not designed to test the effect of TXA on the reduction of PPH incidence, nor on the incidence of rare but severe adverse effects. Large, adequately powered multicenter randomized controlled trials are required before the widespread use of TXA for preventing PPH can be recommended.

The investigators propose a multicentre randomised, double-blind, placebo-controlled trial, with two parallel groups.

Individual information on the trial will be provided to women in late pregnancy during prenatal visits. This information will be repeated when the women arrive in the delivery room; the women then will confirm their participation and provide informed written consent before delivery, when, in the opinion of the investigator, the woman is likely to have a vaginal delivery with a minimum of 4 cm of cervix dilatation.

The intervention will be the intravenous administration of a 10-ml blinded ampoule of the study drug (either 1g TXA or placebo according to the randomisation order), slowly (over 30-60 seconds), within 2 minutes after birth and prophylactic oxytocin administration, and once the cord has been clamped.

All other aspects of management of the third stage will be identical in both arms:

* Routine prophylactic intravenous injection of 5 IU oxytocin at delivery of the anterior shoulder or within 2 minutes after birth
* Placement of a graduated (100 mL graduation) collector bag just after birth, left in place until the birth attendant judges that bleeding has stopped, and always at least for 15 minutes. When a woman is included in the trial, a bag will be prepared and ready to be put in place as soon as the baby is born and placed on the mother's belly; if needed, a second staff person will be present to help in managing both the baby and the bag. This will make it possible to collect and measure vaginal blood loss objectively during the immediate postpartum.
* Manual removal of the placenta at 30 minutes after birth if not expelled in absence of bleeding.
* Rapid suturing of the episiotomy, in accordance with good clinical practices
* Systematic use of uterotonic drugs after third stage of labor is not recommended.
* Controlled cord traction (CCT) will be left at the discretion of the practitioner.

If PPH occurs, standardised management will be provided according to the department's protocol. In particular, the use of TXA for the treatment of PPH will be allowed and left at the discretion of the practitioner according to the department's protocol.

The duration of the participation of each patient included in the trial will be from inclusion through 3 months postpartum.

The planned total duration of the trial will be 34 months including 23 months of patient inclusion

ELIGIBILITY:
Inclusion Criteria:

* Age≥ 18 years
* Planned vaginal delivery
* Term ≥ 35 weeks of gestation
* Singleton pregnancy
* Informed consent form signed

Exclusion Criteria:

* History of venous (deep vein thrombosis and/or pulmonary embolism) or arterial (angina pectoris, myocardial infarction, stroke) thrombosis.
* History of epilepsy or seizure
* Any known cardiovascular, renal, liver disorders
* Auto-immune disease
* Sickle cell disease
* Severe hemorrhagic disease
* Placenta previa
* Abnormally invasive placenta (placenta accreta/increta/percreta)
* Abruptio placentae
* Eclampsia; hemolysis, elevated liver enzymes, low platelet count (HELLP) syndrome
* Multiple pregnancy
* In utero foetal death
* Administration of Low-Molecular-Weight Heparin or antiplatelet agents seven days before delivery
* Poor understanding of the French language

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4079 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Incidence of PPH | 24 hours after birth
  Incidence of PPH defined by blood loss ≥ 500 ml, measured with a graduated collector bag

SECONDARY OUTCOMES:
Mean blood loss at 15 minutes after birth | 15 minutes after birth
  Measured with a collector bag left in place at least 15 minutes to have one measure of blood loss at the same time point in all women
Mean total blood loss | Up to 24 hours after birth
  Measured at collector bag removal
Incidence of severe PPH | 24 hours after birth
  Incidence of PPH defined by blood loss ≥ 1000 ml, measured with a graduated collector bag
Need for supplementary uterotonic treatment | 24 hours after birth
  Proportion of women requiring supplementary uterotonic treatment including sulprostone
Postpartum transfusion | Duration of postpartum hospital stay, an expected average of 3 days
  Proportion of women transfused in postpartum
Need for invasive second-line procedures for PPH | Duration of postpartum hospital stay, an expected average of 3 days
  Any of the following: arterial embolization, pelvic arterial ligation, uterine compression suture, hysterectomy
Hemoglobin peripartum delta | 2 days postpartum
  Mean difference between the hemoglobin values before delivery and on the 2nd day postpartum in the absence of a transfusion of packed red blood cells.
Hematocrit peripartum delta | 2 days postpartum
  Mean difference between the hematocrit values before delivery and on the 2nd day postpartum in the absence of a transfusion of packed red blood cells
Hemodynamic tolerance | 15, 30, 45, 60 and 120 minutes after delivery
  Heart rate, blood pressure
Mild adverse effects | Stay in labor ward, an expected average of 2 hours
  Nausea, vomiting, phosphenes, dizziness
Tolerance lab tests | Day 2 postpartum
  Urea, creatinemia, prothrombin time, active prothrombin time, fibrinogenemia, aspartate and alanine transaminase, total bilirubin
Severe adverse effects | Up to 12 weeks after delivery
  Deep venous thrombosis, pulmonary embolism, myocardial infarction, renal failure needing dialysis

OTHER OUTCOMES:
Women's satisfaction | Day 2 postpartum
  self-questionnaire
Psychological status | 2 months postpartum
  self questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Loic SENTILHES, MD PhD, Principal Investigator — Department of Obstetrics, Angers University Hospital Center; Catherine DENEUX-THARAUX, MD PhD, Study Director — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Angers University Hospital, Angers, France

REFERENCES:
- [Background] Novikova N, Hofmeyr GJ. Tranexamic acid for preventing postpartum haemorrhage. Cochrane Database Syst Rev. 2010 Jul 7;(7):CD007872. doi: 10.1002/14651858.CD007872.pub2. PMID 20614466
- [Background] Peitsidis P, Kadir RA. Antifibrinolytic therapy with tranexamic acid in pregnancy and postpartum. Expert Opin Pharmacother. 2011 Mar;12(4):503-16. doi: 10.1517/14656566.2011.545818. Epub 2011 Feb 4. PMID 21294602
- [Background] Sentilhes L, Daniel V, Darsonval A, Deruelle P, Vardon D, Perrotin F, Le Ray C, Senat MV, Winer N, Maillard F, Deneux-Tharaux C. Study protocol. TRAAP - TRAnexamic Acid for Preventing postpartum hemorrhage after vaginal delivery: a multicenter randomized, double-blind, placebo-controlled trial. BMC Pregnancy Childbirth. 2015 Jun 14;15:135. doi: 10.1186/s12884-015-0573-5. PMID 26071040
- [Background] Sentilhes L, Lasocki S, Ducloy-Bouthors AS, Deruelle P, Dreyfus M, Perrotin F, Goffinet F, Deneux-Tharaux C. Tranexamic acid for the prevention and treatment of postpartum haemorrhage. Br J Anaesth. 2015 Apr;114(4):576-87. doi: 10.1093/bja/aeu448. Epub 2015 Jan 8. PMID 25571934
- [Derived] Sentilhes L, Winer N, Azria E, Senat MV, Le Ray C, Vardon D, Perrotin F, Desbriere R, Fuchs F, Kayem G, Ducarme G, Doret-Dion M, Huissoud C, Bohec C, Deruelle P, Darsonval A, Chretien JM, Seco A, Daniel V, Deneux-Tharaux C; Groupe de Recherche en Obstetrique et Gynecologie. Tranexamic Acid for the Prevention of Blood Loss after Vaginal Delivery. N Engl J Med. 2018 Aug 23;379(8):731-742. doi: 10.1056/NEJMoa1800942. PMID 30134136